CLINICAL TRIAL: NCT00911326
Title: A Ph 3, Prospective, Open-Label, Multicenter Study of Lymphoseek®-Identified Sentinel Lymph Nodes (SLNs) Relative to the Path Status of Non SLN in an Elective Neck Dissection in Cutaneous Head and Neck and Intraoral Squamous Cell Carcinoma
Brief Title: Evaluation of Sentinel Lymph Nodes in Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was terminated early based on an interim review by the Data and Safety Monitoring Committee for positive efficacy outcome and no safety concerns.
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NEO3-06
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lymphoseek — Single injection of 50 micrograms Lymphoseek radiolabeled with either 0.5 mCi (for same day surgery) or 2.0 mCi (for next day surgery) of Tc 99m
  Other Names: Tc-99m Tilmanocept (Lymphoseek)

SUMMARY:
The purpose of this study is to determine the false negative rate (FNR) associated with Lymphoseek-identified sentinel lymph nodes (SLNs) relative to the pathological status of non-sentinel lymph nodes in elective neck dissection (END) in head & neck squamous cell carcinoma (HNSCC). NEO3-06 (this study) is a Phase 3 clinical trial designed to supplement NEO3-05, a completed Phase 3 clinical trial conducted in patients with breast cancer or melanoma. NEO3-05 was designed to establish Lymphoseek as an effective radio-diagnostic agent to be used in the intraoperative localization of lymph tissue (nodes) in the lymphatic pathway draining the primary site of a tumor.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following inclusion criteria by the end of the screening phase should be considered for admission to the study:

1. The patient has provided written informed consent with Health Insurance Portability and Accountability Act (HIPAA) authorization before participating in the study.
2. The patient has a diagnosis of primary squamous cell carcinoma of the head and neck either cutaneous or intra-oral that is anatomically located in: mucosal lip, buccal mucosa, lower alveolar ridge, upper alveolar ridge, retromolar gingiva (retromolar trigone), floor of the mouth, hard palette or oral (mobile) tongue, stage T1-T4a, N0, M0.
3. Clinical nodal staging (N0) has been confirmed by negative results from contrast CT scan or gadolinium-enhanced MRI or lateral and central neck ultrasound. PET scan cannot be used for this evaluation.
4. Imaging of the regional nodal basin has been performed within 30 days of the planned lymphadenectomy.
5. The patient is a candidate for surgical intervention, with intraoperative lymphatic mapping and END included in the surgical plan.
6. Patients with prior malignancy are allowed provided the patient meets the following criteria:

   Underwent potentially curative therapy for all prior malignancies and is deemed low risk for recurrence; AND No malignancy for the past 5 years (except effectively treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix effectively treated with surgery alone, lobular carcinoma in situ of the ipsilateral or contralateral breast treated with surgery alone, or carcinoma of the mouth that is in situ or minimally invasive) and no evidence of recurrence.
7. The patient is at least 18 years of age at the time of consent.
8. The patient has an Eastern Cooperative Oncology Group (ECOG) status of Grade 0 - 2.
9. If the patient is a female, the patient has a confirmed negative pregnancy test within 72 hours priors to administration of Lymphoseek, OR has documentation of surgical sterilization, OR has documented evidence of postmenopausal status for at least 1 year.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria at the end of the screening phase will not be enrolled in the study:

1. The patient has a diagnosis of squamous cell carcinoma of the head and neck in the following anatomical areas: non-mobile base of the tongue, oral pharynx, nasal pharynx, hypo-pharynx and larynx.
2. The patient is pregnant or lactating.
3. The patient has clinical or radiological evidence of metastatic cancer to the regional lymph nodes.
4. Patients with a history of neck dissection, or gross injury to the neck that would preclude reasonable surgical dissection for this study, or radiotherapy to the neck.
5. Patients who have had other nuclear imaging studies conducted within 15 days or consenting.
6. The patient is actively receiving systemic cytotoxic chemotherapy.
7. Patient is currently participating in another investigational drug study or participated within 30 days prior to consenting.
8. Patient is on immunosuppressive or anti-monocyte or immunomodulatory therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie C Abbruzzese, MS RD, Study Director — Navidea Biopharmaceuticals
Locations (13):
- United States (13):
  - University of Alabama, Birmingham, Birminham, Alabama
  - Moores UCSD Cancer Center, La Jolla, California
  - San Diego VA Hospital, San Diego, California
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Mississippi, Jackson, Mississippi
  - University of Missouri-Ellis Fischel Cancer Center, Columbia, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MD Anderson, Houston, Texas

REFERENCES:
- [Derived] Agrawal A, Civantos FJ, Brumund KT, Chepeha DB, Hall NC, Carroll WR, Smith RB, Zitsch RP, Lee WT, Shnayder Y, Cognetti DM, Pitman KT, King DW, Christman LA, Lai SY. [(99m)Tc]Tilmanocept Accurately Detects Sentinel Lymph Nodes and Predicts Node Pathology Status in Patients with Oral Squamous Cell Carcinoma of the Head and Neck: Results of a Phase III Multi-institutional Trial. Ann Surg Oncol. 2015 Oct;22(11):3708-15. doi: 10.1245/s10434-015-4382-x. Epub 2015 Feb 11. PMID 25670018
- [Derived] Marcinow AM, Hall N, Byrum E, Teknos TN, Old MO, Agrawal A. Use of a novel receptor-targeted (CD206) radiotracer, 99mTc-tilmanocept, and SPECT/CT for sentinel lymph node detection in oral cavity squamous cell carcinoma: initial institutional report in an ongoing phase 3 study. JAMA Otolaryngol Head Neck Surg. 2013 Sep;139(9):895-902. doi: 10.1001/jamaoto.2013.4239. PMID 24051744

RESULTS

PARTICIPANT FLOW:
Groups:
- Lymphoseek: Intraoral and cutaneous (head and neck) squamous cell carcinoma (T1-T4, N0, M0) patients to receive a single dose of 50 µg Lymphoseek radiolabeled with 0.5 or 2.0 mCi Tc 99m for sentinel lymph node biopsy and elective neck dissection of cervical lymph nodes.
Period: Overall Study
Arm/Group | Lymphoseek
Started | 101
Completed | 85
Not Completed | 16

BASELINE CHARACTERISTICS:
Population: Of the 101 participants who enrolled in the trial, 85 were administered the study agent, Lymphoseek, and therefore this participant number is used for the baseline analysis.
Groups:
- Lymphoseek: Enrolled patients who were administered any injection of Lymphoseek.
Arm/Group | Lymphoseek
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 64
Region of Enrollment [Number; unit: participants]
  United States | 85
Clinical tumor stage [Number; unit: participants] — From the American Joint Committee on Cancer, Manual for Staging of Cancer 6th Edition.
  T1: tumor 2 cm or less in greatest dimension; T2: tumor more than 2 cm but not more than 4 cm (for lip and oral cavity SCC) or 5 cm (for cutaneous SCC) in greatest dimension; T3: tumor more than 4 cm (for lip and oral cavity SCC) or 5 cm (for cutaneous SCC) in greatest dimension; T4: tumor invades adjacent structures (for lip and oral cavity SCC) or deep extradermal structures (for cutaneous SCC).
  participants
    T1 | 26
    T2 | 46
    T3 | 7
    T4 | 6
Tumor location [Number; unit: participants]
  Buccal mucosa | 8
  Cutaneous | 6
  Floor of the mouth | 20
  Lower alveolar ridge | 3
  Mucosal lip | 1
  Oral tongue | 43
  Retromolar gingiva | 4

OUTCOME MEASURES:

1. Primary Outcome: False Negative Rate (FNR)
Description: The FNR is calculated as a percentage from the ratio of false negatives to the sum of true positives plus false negatives. The FNR point estimate was the observed rate and was made on a per-patient basis relative to patients with pathology-positive nodes.
Time Frame: Surgery after injection of Lymphoseek
Measure: Number (95% Confidence Interval); unit: % of pathology-positive participants
Groups:
- Intent-to-treat (ITT): All enrolled patients who were injected with Lymphoseek, who underwent surgery, and had at least one lymph node removed (sentinel or non-sentinel) for which the pathology status (presence/absence of tumor cells) was confirmed.
Arm/Group | Intent-to-treat (ITT)
Number analyzed (Participants) | 83
% of pathology-positive participants | 2.56 [0.06 to 13.49]

2. Secondary Outcome: Negative Predictive Value (NPV)
Description: The NPV is calculated as a percentage from the ratio of true negatives to the sum of true negatives plus false negatives. The NPV point estimate was the observed rate and was made on a per-patient basis relative to patients predicted to be pathology-negative.
Time Frame: Surgery after injection of Lymphoseek
Measure: Number (95% Confidence Interval); unit: % of participants predicted negative
Arm/Group | Intent-to-treat (ITT)
Number analyzed (Participants) | 83
% of participants predicted negative | 97.8 [88.2 to 99.9]

3. Secondary Outcome: Overall Accuracy
Description: The overall accuracy is calculated as a percentage from the ratio of (true positives + true negatives) / (true positives + false negatives + true negatives). The overall accuracy point estimate was the observed rate and was made on a per-patient basis relative to all patients in the intent-to-treat population.
Time Frame: Surgery after injection of Lymphoseek
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intent-to-treat (ITT)
Number analyzed (Participants) | 83
percentage of participants | 98.8 [93.5 to 99.9]

4. Secondary Outcome: Lymph Node Detection Rate
Description: The rate of the subjects for whom Lymphoseek identified at least 1 sentinel lymph node. The detection rate point estimate was the observed rate and was made on a per-patient basis relative to all patients in the intent-to-treat population.
Time Frame: Surgery after injection of Lymphoseek
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intent-to-treat (ITT)
Number analyzed (Participants) | 83
percentage of participants | 97.6 [91.6 to 99.7]

ADVERSE EVENTS:
Time Frame: Overall study
Arm/Group | Lymphoseek
Serious Adverse Events (participants affected / at risk) | 11/85
Other Adverse Events (participants affected / at risk) | 6/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lymphoseek (N=85)
Atrial fibrillation (Cardiac disorders) | 1 — Not related to Lymphoseek.
Mouth haemorrhage (Gastrointestinal disorders) | 1 — Not related to Lymphoseek.
Salivary gland fistula (Gastrointestinal disorders) | 1 — Not related to Lymphoseek.
Post procedural infection (Infections and infestations) | 2 — Not related to Lymphoseek.
Arterial injury (Injury, poisoning and procedural complications) | 1 — Not related to Lymphoseek.
Presyncope (Nervous system disorders) | 1 — Not related to Lymphoseek.
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 — Not related to Lymphoseek.
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 — Not related to Lymphoseek.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 — Not related to Lymphoseek.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 — Not related to Lymphoseek.
Haematoma (Vascular disorders) | 1 — Not related to Lymphoseek.
Hypotension (Vascular disorders) | 1 — Not related to Lymphoseek.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lymphoseek (N=85)
Diarrhoea (Gastrointestinal disorders) | 6 — Not related to Lymphoseek.

LIMITATIONS AND CAVEATS:
The study was prospectively structured to include an interim analysis at 33.3% enrollment. The trial was terminated early based on an interim review by the Data and Safety Monitoring Committee for positive efficacy outcome and lack of safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not submit a publication to journals or professional societies without the prior written approval of the Sponsor.